CLINICAL TRIAL: NCT03380546
Title: Non-inferiority Between Acarbose and Prandial Insulin for the Treatment of Gestational Diabetes Mellitus: a Randomized Multicenter and Prospective Trial. ACARB-GDM Study.
Brief Title: Acarbose and Prandial Insulin for the Treatment of Gestational Diabetes Mellitus.
Acronym: ACARB-GDM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficulty in recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P150942
Record Dates: First submitted 2017-11-07; First posted 2017-12-21 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: Diabetes; Pregnancy; Gestational; Acarbose
MeSH Terms: conditions — Diabetes Mellitus | interventions — Acarbose; Insulin, Short-Acting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- acarbose (Experimental): The women will receive acarbose with a progressive increase of dose according to post prandial glucose values and digestive tolerance, with a maximal dose of 3 x 100 mg /day
  Interventions: Drug: Acarbose
- prandial insulin (Active Comparator): The women will receive prandial insulin according to usual practice (routine care according to French recommendations): before each meal, with dose titration according to post prandial values.
  Interventions: Drug: Prandial insulin

INTERVENTIONS:
Drug: Acarbose — Women will receive acarbose at an initial dose of 50 mg once daily in the beginning of the meal for which the postprandial glucose value is the highest, with progressive increase every 2 days or more: adding a pill before another meal, and then increasing dose of acarbose to 100 mg if post-prandial glucose goals are not obtained, with a maximal dose of 3 x 100 mg / day.
  Other Names: Glucor 50 mg
  Arms: acarbose
Drug: Prandial insulin — Women will receive prandial fast-acting insulin according to usual practice (routine care according to French recommendations), i.e. one injection before each meal usually.
  Other Names: Rapid acting insulin analog
  Arms: prandial insulin

SUMMARY:
Caring for women with gestational diabetes mellitus (GDM) is very time-consuming. Therapeutic strategy includes dietary and lifestyle measures and additional insulin therapy for 15 to 40% of the women with GDM if the glycemic targets are not achieved after a period of 1 to 2 weeks of diet. Insulin therapy is imperfect for the following main reasons: need for education (i.e. subcutaneous administration, dose titration), hypoglycemia and weight gain, limited acceptance and high cost. Psychosocial deprivation is associated with more cases of GDM and health accessibility may be unequal.

Glucosidase inhibitors (acarbose) reduce intestinal absorption of starch and reduce the rate of complex carbohydrate digestion. It mainly lowers postprandial glucose values and is used in type 2 diabetes for a long time. Less than 2% of a dose is absorbed as active drug in adults, with 34% of the metabolites found in the systemic circulation. Doses of up to 9 and 32 times the human dose were not teratogenic in pregnant rats or rabbits. Limited but reassuring data during pregnancy are available. Acarbose was well tolerated (little gestational weight gain, no hypoglycemia) with digestive discomfort in some women, balanced by treatment satisfaction as compared with insulin injections. Our hypothesis is that treatment aiming to control postprandial glucose values with acarbose as compared with prandial insulin injection will be as efficient and safe, but more convenient and less expensive.

DETAILED DESCRIPTION:
Phase III study. Prospective, multicenter, non-inferiority, randomized, open-labelled and controlled study with two arms.

1. In the 37 participating hospitals: selection of women with GDM who have unmet post prandial glycemic targets between 14 and 37 (+6 days) weeks of amenorrhea after at least 7 days of dietary and lifestyle measures. They may be treated with basal insulin to control pre prandial glucose values.
2. Explanation of protocol, with signature of consent in case of acceptation.
3. Randomization

   . Experimental group: The women will receive acarbose with a progressive increase of dose according to post prandial glucose values and digestive tolerance, with a maximal dose of 3 x 100 mg / day. The progressive titration of acarbose reduces gastro-intestinal side effects.

   Patients who have not reached the glycemic targets at this highest tolerated dose for at least one meal will receive instead prandial insulin therapy for each meal, whereas acarbose will be stopped. Failure to reach post-prandial target will be defined as 3 or more post-prandial glycaemic values ≥ 1.20 g/L for a given meal in a week (3 values out of 7) after the two weeks of dose adjustment.

   · Control group: The women will receive prandial insulin according to usual practice (routine care according to French recommendations): before each meal, with dose titration according to post prandial values.

   Basal insulin may be necessary in both arms to control pre-prandial glucose values.

   At delivery:

   - Maternal blood samples : 14 ml of blood will be collected at the same time as the sample routinely collected just before delivery for irregular agglutinin test measurement, when the women are perfused.

   - Cord fluid : 7 ml will be collected at the same as cord fluid pH is routinely measured just after delivery. There will be 5 aliquots to prepare.

   The aliquots previously labelled and stowed in the specific boxes for the study will be stored locally and will be transported to the "Centre de Ressources Biologiques"(CRB) of the Jean Verdier Hospital.
4. Routine monitoring of the women with GDM in both arms, up to delivery. No use of other oral hypoglycemic agents during pregnancy.
5. Last consultation three months after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Singleton pregnancy
* GDM diagnosed during pregnancy according to IADPSG criteria
* Self-monitoring of blood glucose
* After at least 7 days of dietary and lifestyle measures, unreached post-prandial glucose control
* 14-37 (+ 6 days) amenorrhea weeks at the time of randomization
* Signed informed consent

Exclusion Criteria:

* Prandial insulin use before randomization during this pregnancy
* Use of other oral hypoglycemic agents during this pregnancy
* Multiple pregnancy
* Known hepatic insufficiency
* Long time corticosteroid treatment
* Pre-existing diabetes in pregnancy
* Overt diabetes diagnosed during pregnancy (IADPSG criteria)
* Lack of Social Insurance
* Insufficient understanding
* Participant in another investigational drug study at inclusion visit
* Contraindications of acarbose
* Fetal malformation diagnosed by previous fetal ultrasound

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The participants in this study are pregnant women with gestational diabetes mellitus.
Enrollment: 341 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Composite endpoint: birth weight ≥ 90th percentile for gestational age (large for gestational age: LGA) and/or neonatal hypoglycemia and/or shoulder dystocia and/or birth injury. | At delivery
  LGA defined as birth weight greater than the 90th percentile for a standard French population
  * Neonatal hypoglycemia defined as at least a blood glucose value less than a 2.0 mmol/l during the two first days of life;
  * Shoulder dystocia, defined as vaginal cephalic delivery that requires additional obstetric manoeuvres to deliver the fetus after the head has delivered and gentle traction has failed. We will only consider rotational maneuvers such as Rubin II or Woods corkscrew or Jaquemier maneuvers
  * Birth injury defined as plexus injury or clavicle fracture.

SECONDARY OUTCOMES:
GLUCOSE CONTROL: Capillary glucose levels | From two weeks after inclusion : 14 and 37 (+6 days) weeks of amenorrhea to delivery
  The women will be asked to perform 6 measures a day. Capillary glucose values will be retrieved from the glucose meter, and if not available, from the woman's diary.
GLUCOSE CONTROL: HbA1c | At delivery
  Centralized measurement
GLUCOSE CONTROL: Need for and dose/day of basal and prandial insulin in both arms | At delivery
  This information will be retrieved from the glucose meter, and if not available, from the woman's diary.
Neonatal complications : Birth weight and height, | At delivery
  Birth weight ≥ 4000g Birth weight ≥ 4500g
Neonatal complications : Small for gestational age infant | At delivery
  SGA: birth weight lower than the 10th percentile for a standard French population
Maternal complications : Preeclampsia | From two weeks after inclusion to delivery
  Preeclampsia (blood pressure ≥ 140/90 mmHg on two measurements four hours apart and proteinuria of at least 300 mg/24 hours or 3+ or more on dipstick testing or proteinuria/creatininuria >30 in a random urine sample).
Maternal complications : Pregnancy-induced hypertension | From two weeks after inclusion : 14 and 37 (+6 days) weeks of amenorrhea to delivery
  In women with no known hypertension before pregnancy, blood pressure ≥ 140/90 mmHg on two measurements four hours apart without proteinuria and having needed to begin anti-hypertensive therapy
Neonatal complications : Preterm delivery | At delivery
  * Late preterm infant (between 32 and 37 completed weeks' gestation)
  * Very preterm infant (28-31 completed weeks' gestation)
  * Extreme preterm infant (less than 28 completed weeks' gestation)
Neonatal complications : Low Apgar score | At delivery
  5-min Apgar score < 7
Neonatal complications : Neonatal respiratory distress syndrome | At delivery
  based on the clinical course, chest X-ray finding, blood gas and acid-base values
Neonatal complications : Intrauterine fetal or neonatal death; | From two weeks after inclusion to delivery
  These endpoints will be extracted from the women' charts
Acceptance/satisfaction of two strategies : -Quality of life -Satisfaction questionnaires | At delivery
  Medical Outcomes Study 36-Item Short-Form General Health Survey (SF-36)
  - use of analogic scales
Side effects of drugs : Maternal hypoglycemia | during the 7 months of treatment
  * Severe hypoglycemia: requiring assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma/capillary glucose to normal is considered sufficient evidence that the event was induced by a low plasma/capillary glucose concentration.
  * event during which typical symptoms of hypoglycemia are accompanied by a measured capillary glucose concentration <70 mg/dL (<3.9 mmol/L).
  * Asymptomatic hypoglycemia: event not accompanied by typical symptoms of hypoglycemia but with a measured capillary glucose concentration <60 mg/dL (<3.3 mmol/L).
Gastro-intestinal side effects | from two weeks after inclusion : 14 to 36 weeks of gestation to delivery
  The events occuring during the last 14 days of pregnancy or gastro-intestinal side effects leading to treatment withdrawl
Results of oral glucose tolerance test and HbA1c measurement | 3 months after delivery
  Test will be performed by the women before follow up visit
Infant anthropometrics. | At month 1, month 2 and month 3
  These data will be collected from children's health record
Conservation of serum and plasma; cord fluid. The samples may be used for further analyses ancillary studies and which could be beneficial for GDM care based on evolution in scientific knowledge. | within 10 years after the end of the study
  * The blood samples will be collected at the same time as the sample routinely collected just before delivery for irregular agglutinin test measurement.
  * Cord fluid will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COSSON, MD-PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Jean Verdier Hospital, Bondy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rowan JA, Hague WM, Gao W, Battin MR, Moore MP; MiG Trial Investigators. Metformin versus insulin for the treatment of gestational diabetes. N Engl J Med. 2008 May 8;358(19):2003-15. doi: 10.1056/NEJMoa0707193. PMID 18463376
- [Background] Langer O, Conway DL, Berkus MD, Xenakis EM, Gonzales O. A comparison of glyburide and insulin in women with gestational diabetes mellitus. N Engl J Med. 2000 Oct 19;343(16):1134-8. doi: 10.1056/NEJM200010193431601. PMID 11036118
- [Background] Holt RI, Lambert KD. The use of oral hypoglycaemic agents in pregnancy. Diabet Med. 2014 Mar;31(3):282-91. doi: 10.1111/dme.12376. PMID 24528229
- [Background] Zarate A, Ochoa R, Hernandez M, Basurto L. [Effectiveness of acarbose in the control of glucose tolerance worsening in pregnancy]. Ginecol Obstet Mex. 2000 Jan;68:42-5. Spanish. PMID 10774102
- [Background] Platt J, O'Brien W. Title Acarbose therapy for gestational diabetes: a retrospective cohort study (abstract). Review AJOG 2003;189:S107